CLINICAL TRIAL: NCT02684305
Title: Stepwise Labor Induction Following Failure of Prostaglandin Vaginal Insert for Labor Induction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 686-15- TLV
Record Dates: First submitted 2016-01-28; First posted 2016-02-17 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Induction of Labor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Administration of Propess (Experimental): All women who failed induction of labor using vaginal insert slow release of dinoprostone 10 mg (Propess), defined as bishop score ≤ 7 24 hours after propess insertion will be randomized to one of the following treatment arms:
  1.Administration of Propess for additional 24 hours.
  Interventions: Drug: Administration of Propess
- Intravenous oxytocin infusion + balloon (Experimental): All women who failed induction of labor using vaginal insert slow release of dinoprostone 10 mg (Propess), defined as bishop score ≤ 7 24 hours after propess insertion will be randomized to one of the following treatment arms:
  2. Intravenous oxytocin infusion combined with intracervical balloon administration, inflated with 60cc of saline.
  Interventions: Device: balloon; Drug: Intravenous oxytocin infusion

INTERVENTIONS:
Drug: Administration of Propess — 1. History taking and physical examination including cervical length
  2. Eligibility assessment
  3. Explanation regarding the study protocol
  4. Signed informed consent (at VAS<3)
  5. Women agreeing to continued induction of labor 24 hours after insertion of Propess, will be randomized using sealed envelopes to the subsequent method of induction of labor (additional vaginal insert vs. oxytocin infusion with intracervical balloon insertion with 60ml saline). Treatment will be given according to the pre-existing and approved departmental protocol. The protocol for oxytocin infusion is 4 units of Pitocin in 10 cc 0.9% NaCl, infused at a rate of 0.4 ml/hour. Infusion rate will be increased every 20 minutes until 3-4 contractions every 10 minutes are produced.
  Follow up on all women will be performed from the time of second agent induction until discharge from hospital postpartum.
  Arms: Administration of Propess
Device: balloon — 1. History taking and physical examination including cervical length
  2. Eligibility assessment
  3. Explanation regarding the study protocol
  4. Signed informed consent (at VAS<3)
  5. Women agreeing to continued induction of labor 24 hours after insertion of Propess, will be randomized using sealed envelopes to the subsequent method of induction of labor (additional vaginal insert vs. oxytocin infusion with intracervical balloon insertion with 60ml saline). Treatment will be given according to the pre-existing and approved departmental protocol. The protocol for oxytocin infusion is 4 units of Pitocin in 10 cc 0.9% NaCl, infused at a rate of 0.4 ml/hour. Infusion rate will be increased every 20 minutes until 3-4 contractions every 10 minutes are produced.
  Follow up on all women will be performed from the time of second agent induction until discharge from hospital postpartum.
  Arms: Intravenous oxytocin infusion + balloon
Drug: Intravenous oxytocin infusion — 1. History taking and physical examination including cervical length
  2. Eligibility assessment
  3. Explanation regarding the study protocol
  4. Signed informed consent (at VAS<3)
  5. Women agreeing to continued induction of labor 24 hours after insertion of Propess, will be randomized using sealed envelopes to the subsequent method of induction of labor (additional vaginal insert vs. oxytocin infusion with intracervical balloon insertion with 60ml saline). Treatment will be given according to the pre-existing and approved departmental protocol. The protocol for oxytocin infusion is 4 units of Pitocin in 10 cc 0.9% NaCl, infused at a rate of 0.4 ml/hour. Infusion rate will be increased every 20 minutes until 3-4 contractions every 10 minutes are produced.
  Follow up on all women will be performed from the time of second agent induction until discharge from hospital postpartum.
  Arms: Intravenous oxytocin infusion + balloon

SUMMARY:
Induction of labor is one of the most common obstetrical medical procedures performed today. Iatrogenic stimulation of uterine contractions prior to the onset of spontaneous labor is undertaken for various maternal and fetal indications and spans 20% of deliveries today.

1. During the past years there has been an additional rise due to elective inductions
2. Induction is undertaken when potential risks of prolonging pregnancy outweigh the risks of induced delivery, particularly those associated with post-term pregnancy, rupture of membranes, oligohydramnios and additional fetal and maternal conditions that pose risks to mother and fetus.

In many circumstances of women with an unfavorable cervix (Bishop score of 7 or less) sequential induction with more than one agent is necessary. To date, no trial has compared the optimal subsequent ripening method after the preliminary use of dinoprostone (prostaglandin E2). In this trial investigators aim to compare the obstetrical outcomes of subsequent induction in women admitted for induction of labor with Bishop score <7 or less 24 hours after the insertion of vaginal prostaglandin insert (Propess). Two methods of routine induction of labor will be compared: An additional Propess induction for another 24 hours vs. intravenous oxytocin infusion combined with intra-cervical balloon insertion.

DETAILED DESCRIPTION:
Induction of labor is one of the most common obstetrical medical procedures performed today. Iatrogenic stimulation of uterine contractions prior to the onset of spontaneous labor is undertaken for various maternal and fetal indications and spans 20% of deliveries today

1. During the past years there has been an additional rise due to elective inductions
2. Induction is undertaken when potential risks of prolonging pregnancy outweigh the risks of induced delivery, particularly those associated with post-term pregnancy, rupture of membranes, oligohydramnios and additional fetal and maternal conditions that pose risks to mother and fetus.

In many circumstances of women with an unfavorable cervix (Bishop score of 7 or less) sequential induction with more than one agent is necessary. To date, no trial has compared the optimal subsequent ripening method after the preliminary use of dinoprostone (prostaglandin E2). In this trial investigators aim to compare the obstetrical outcomes of subsequent induction in women admitted for induction of labor with Bishop score <7 or less 24 hours after the insertion of vaginal prostaglandin insert (Propess). Two methods of routine induction of labor will be compared: An additional Propess induction for another 24 hours vs. intravenous oxytocin infusion combined with intra-cervical balloon insertion.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal age of 18 years or greater
2. Singleton gestation
3. Bishop score of 7 or less 24 hours after the insertion of Propess
4. Pregnancies at 36+0/7 weeks of gestation and beyond
5. Normal fetal heart rate tracings and normal sonogram at admission (ie Vertex, appropriate for gestational age, biophysical score of 8/8, normal amniotic fluid index)
6. No contraindication for prolongation of pregnancy (e.g. intrauterine infection, placental abruption, etc.)

Exclusion Criteria:

1. Situations preventing continuation of induction process in any arm - patient refusal, maternal of fetal conditions necessitating prompt delivery.
2. Rupture of membranes (ROM) after initial Propess insertion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Time from second agent induction to delivery | 48 hours
  Time from second agent induction to active labor

SECONDARY OUTCOMES:
Rate of failed induction defined as 5 cm dilatation | 48 hours
  Defined as 5 cm dilatation with regular contractions
Rate of failed induction defined as regular contractions | 48 hours
  Rate of failed induction defined as regular contractions (over 3 contractions in 30 min)
cesarean sections rate | 48 hours
  Number of cesarean sections rate due to tachysystole and non-reassuring fetal heart rate.

CONTACTS AND LOCATIONS:
Overall Officials: yariv yogev, professor, Principal Investigator — Tel Aviv Medical Center

IPD SHARING:
Plan to Share IPD: No